CLINICAL TRIAL: NCT01297452
Title: A Phase I Study of BKM120 + Carboplatin + Paclitaxel for Patients With Advanced Solid Tumors
Brief Title: BKM120 + Carboplatin + Paclitaxel for Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Sai Life Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-192
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Solid Tumors
Keywords: BKM120; CARBOPLATIN; TAXOL (PACLITAXEL); Chemotherapy; 10-192
MeSH Terms: interventions — Paclitaxel; Carboplatin; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BKM120 (days 1 - 21) + paclitaxel + carboplatin (Experimental): This will be a single institution phase I study. The primary objectives are to determine the maximum tolerated dose of BKM120 administered with paclitaxel + carboplatin on both a 21-day cycle with growth factor support (Group 1)
  Interventions: Drug: BKM120 days 1 - 21 plus paclitaxel + carboplatin; Drug: BKM120, Paclitaxel + Carboplatin
- BKM120 (days 1 - 28, ) + paclitaxel + carboplatin (Experimental): This will be a single institution phase I study. The primary objectives are to determine the maximum tolerated dose of BKM120 administered + paclitaxel with carboplatin on a 28-day cycle with growth factor support and a 28-day cycle (Group 2).
  Interventions: Drug: BKM120 (days 1 - 28, ) plus paclitaxel + carboplatin
- BKM120 (days 1-21) + paclitaxel (day 1) + carboplatin (day 1) (Experimental): EXPANSION COHORT A BKM120 100 mg (days 1 - 21, per dose escalation scheme) plus paclitaxel (200 mg/m2 intravenously, day 1) + carboplatin (AUC 6 intravenously, day 1) on a 21-day cycle. After enrollment to Groups 1 and 2 has been completed and all patients in Group 1 and 2 have completed the DLT monitoring period, up to 6 additional patients will be enrolled in this EXPANSION COHORT A.
  Interventions: Drug: BKM120 (days 1-21) + paclitaxel (day 1) + carboplatin (day 1)
- BKM120 (days 1 - 21) + paclitaxel + carboplatin exp B (Experimental): Expansion Cohort B will be restricted to patients with tumors known to harbor PTEN mutation or homozygous deletion. The regimen in Expansion Cohort B will be the same regimen established in Group 1 of the protocol, with BKM120 (now called buparlisib) at 100 mg/day per oral + paclitaxel (175 mg/m2) + carboplatin (AUC 5), both given intravenously (IV) on day 1 of a 21-day cycle
  Interventions: Drug: BKM120 (days 1 - 28, ) plus paclitaxel + carboplatin

INTERVENTIONS:
Drug: BKM120 days 1 - 21 plus paclitaxel + carboplatin — Patients will receive oral daily BKM120 (days 1 - 21, per dose escalation scheme) plus paclitaxel (175 mg/m2 intravenously, day 1) + carboplatin (AUC 5 intravenously, day 1)on a 21-day cycle. Pegfilgrastim (6 mg/subcutaneously) will be administered on day 2 of each cycle.
  Arms: BKM120 (days 1 - 21) + paclitaxel + carboplatin
Drug: BKM120 (days 1 - 28, ) plus paclitaxel + carboplatin — Patients will receive oral daily BKM120 (days 1 - 28, per dose escalation scheme) plus paclitaxel (80 mg/m2 intravenously, days 1, 8 and 15) + carboplatin (AUC 5 intravenously, day 1) on a 28-day cycle.
  Arms: BKM120 (days 1 - 21) + paclitaxel + carboplatin exp B; BKM120 (days 1 - 28, ) + paclitaxel + carboplatin
Drug: BKM120 (days 1-21) + paclitaxel (day 1) + carboplatin (day 1) — BKM120 100 mg (days 1 - 21, per dose escalation scheme) plus paclitaxel (200 mg/m2 intravenously, day 1) + carboplatin (AUC 6 intravenously, day 1) on a 21-day cycle. After enrollment to Groups 1 and 2 has been completed and all patients in Group 1 and 2 have completed the DLT monitoring period, up to 6 additional patients will be enrolled in this EXPANSION COHORT.A
  Arms: BKM120 (days 1-21) + paclitaxel (day 1) + carboplatin (day 1)
Drug: BKM120, Paclitaxel + Carboplatin — BKM120 100 mg per oral, days 1 - 21 Paclitaxel (175 mg/m2) intravenously on Day 1 Carboplatin (AUC 5) intravenously on Day 1 EXPANSION COHORT B
  Arms: BKM120 (days 1 - 21) + paclitaxel + carboplatin

SUMMARY:
The purpose of this study is to find out the good and bad effects that occur when BKM120 is added to standard chemotherapy with carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed recurrent or metastatic advanced solid tumor, for which there is no curative-intent treatment option. Pathology confirmation must be performed at MSKCC.
* Age ≥ 18 years
* ECOG performance status ≤ 1
* Life expectancy of ≥ 12 weeks
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hemoglobin > 9 g/dL
* Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
* Magnesium ≥ the lower limit of normal
* Adequate liver function.
* Serum bilirubin must be within the upper limit of normal. (ULN). AST and ALT and Alkaline Phosphatase must be within the range allowing for eligibility. In determining eligibility the more abnormal of the two values (AST or ALT) should be used.
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 55 mL/min
* Fasting plasma glucose (FPG) ≤120 mg/dL or ≤6.7 mmol/L
* HbA1c ≤ 8%
* Negative serum pregnancy test within 14 days before starting study treatment in women with childbearing potential
* Ability to swallow oral medication
* EXPANSION COHORT B ONLY: Documented genetic alteration (mutation or homozygous deletion) in the PTEN gene, identified by the MSKCC IMPACT assay platform or other CLIA-approved test.

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor.
* Patients with a known hypersensitivity to BKM120 or to its excipients
* Patients with untreated brain metastases are excluded. However, patients with metastatic CNS tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (incl. radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy
* Patients with acute or chronic liver, renal disease or pancreatitis
* Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as result of patient's mood assessment questionnaire:

  * medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)

    *≥ CTCAE grade 3 anxiety
  * At screening, mood rating scores of ≥ 10 on PHQ-9 and/or ≥ 15 on GAD-7, unless overruled by psychiatrist's assessment
* Patient selects a response of "1, 2, or 3" for question 9 on PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9) Note: The psychiatric judgment overrules the mood assessment questionnaire result/investigators judgment. If mood rating scores do not meet eligibility criteria and/or the investigator deems that a patient has mood disorder that renders the patient ineligible, that patient may not be registered to the study unless there is a subsequent psychiatric clinic consultation in which the psychiatrist overrules the mood assessment questionnaire result/investigator judgment.
* Patients with diarrhea ≥ CTCAE grade 2
* Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:
* ST depression or elevation of ≥ 1.5 mm in 2 or more leads
* Congenital long QT syndrome
* History or presence of sustained ventricular arrhythmias or atrial fibrillation
* Clinically significant resting bradycardia (< 50 beats per minutes) QTc > 480 msec on screening ECG
* Complete left bundle branch block
* Right bundle branch block + left anterior hemiblock (bifascicular block)
* Unstable angina pectoris ≤ 6 months prior to starting study drug
* Acute myocardial infarction ≤ 6 months prior to starting study drug
* Other clinically significant heart disease such as congestive heart failure requiring treatment (NYHA Class III or IV) or uncontrolled hypertension (please refer to WHO-ISH guidelines)
* Patients with uncontrolled diabetes mellitus
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who are currently receiving treatment with QT prolonging medication with a known risk to induce Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to Appendix E for a list of prohibited drugs.
* Patient is currently being treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Appendix B for a list of prohibited CYP 3A4 inhibitors and inducers.
* Patients who have received systemic corticosteroids ≤ 2 weeks prior to starting study drug. Systemic corticosteroids should not be administered with BKM120 (Usage of steroids as premedications and anti-emetics for paclitaxel and carboplatin, per MSKCC guidelines, is allowed). Steroids given as part of pre-medications for imaging studies are not exclusionary.).
* Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy (except alopecia)
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy (except alopecia)
* Patients who have received radiotherapy within ≤ 4 weeks prior to registration
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
* Patient is currently being treated with olanzapine and/or other drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator
* More than 2 prior cytotoxic chemotherapy regimens for recurrent or metastatic disease
* Patients with multifocal peripheral sensory alterations or paresthesias (including tingling) interfering with function, per patient report (example: activities of daily living).
* Patients receiving other investigational therapies
* Patients receiving herbal preparations/medications
* Patients with any prior history of whole pelvic radiation therapy (WPRT)
* EXPANSION COHORT A ONLY: More than one prior cytotoxic chemotherapy regimen (in the setting of recurrent and/or metastatic disease (cytotoxic chemotherapy given as part of neo-adjuvant therapy, adjuvant therapy, or concurrent chemoradiation for curative intent is not included in this exclusion item). This does not apply to Expansion Cohort B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
To establish the phase II recommended dose of daily oral BKM120 | 2 years
  for patients with advanced solid tumors, BKM120 in combination with two different schedules of paclitaxel and carboplatin.
EXPANSION COHORT A:To evaluate the safety and tolerability of daily oral BKM120 (100 mg) + paclitaxel (200 mg/m2) + carboplatin (AUC 6), both given intravenously (IV) on day 1 of a 21-day cycle, with pegfilgrastim support | 2 years
EXPANSION COHORT B: To obtain a preliminary description of efficacy of the regimen established in Group 1 among patients with tumors harboring PTEN mutation or homozygous deletion. | 2 years

SECONDARY OUTCOMES:
To describe the safety of BKM120 combined with paclitaxel and carboplatin, | weekly clinic visits during Cycle 1, on Day 1 of subsequent cycles,
  Patients will be evaluated by MD at weekly clinic visits during Cycle 1, on Day 1 of subsequent cycles, and will have additional evaluations if clinically indicated. Toxicities will be assessed according to NCI common toxicity criteria (CTC) version 4.0
To determine the pharmacokinetic profile of daily BKM120. | 2 years
  when given in combination with carboplatin and paclitaxel. The area under the curve (AUC0→∞), half-life (t½), and maximum concentration (Cmax) for BKM120 will be determined by noncompartmental analysis.(except for Expansion Cohort B)
To describe and tabulate the radiographic response rate of BKM120 in combination with carboplatin and paclitaxel, | 2 years
  there is insufficient sample size to support a formal analysis of response rate. As such, radiographic response data will be tabulated and presented in descriptive form.
Correlative Tissue Studies | 2 years
  we will calculate the proportion of cases with positive staining of PTEN along with a 95% confidence interval, using the Clopper and Pearson method for exact small sample inference. For Sequenom Analysis, we will calculate the proportion of cases that are positive for each mutation

CONTACTS AND LOCATIONS:
Overall Officials: David Hyman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Smyth LM, Monson KR, Jhaveri K, Drilon A, Li BT, Abida W, Iyer G, Gerecitano JF, Gounder M, Harding JJ, Voss MH, Makker V, Ho AL, Razavi P, Iasonos A, Bialer P, Lacouture ME, Teitcher JB, Erinjeri JP, Katabi N, Fury MG, Hyman DM. A phase 1b dose expansion study of the pan-class I PI3K inhibitor buparlisib (BKM120) plus carboplatin and paclitaxel in PTEN deficient tumors and with dose intensified carboplatin and paclitaxel. Invest New Drugs. 2017 Dec;35(6):742-750. doi: 10.1007/s10637-017-0445-0. Epub 2017 Mar 9. PMID 28281183
- [Derived] Hyman DM, Snyder AE, Carvajal RD, Gerecitano JF, Voss MH, Ho AL, Konner J, Winkelmann JL, Stasi MA, Monson KR, Iasonos A, Spriggs DR, Bialer P, Lacouture ME, Teitcher JB, Katabi N, Fury MG. Parallel phase Ib studies of two schedules of buparlisib (BKM120) plus carboplatin and paclitaxel (q21 days or q28 days) for patients with advanced solid tumors. Cancer Chemother Pharmacol. 2015 Apr;75(4):747-55. doi: 10.1007/s00280-015-2693-z. Epub 2015 Feb 12. PMID 25672916
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm